CLINICAL TRIAL: NCT01772680
Title: Zinc and Diabetes in Patients With Thalassemia: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2012-071
Record Dates: First submitted 2013-01-17; First posted 2013-01-21 (Estimated); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Thalassemia
Keywords: Thalassemia; Diabetes; Zinc; Iron-Overload
MeSH Terms: conditions — Thalassemia; Diabetes Mellitus; Iron Overload

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Zinc Supplementation (Experimental): 25 mg elemental Zinc as Zn sulfate in capsule form taken daily for 3 months
  Interventions: Dietary Supplement: Zinc Supplementation

INTERVENTIONS:
Dietary Supplement: Zinc Supplementation — 25 mg elemental zinc taken as zinc sulfate in capsule form taken daily for 3 months

SUMMARY:
The primary aim of this study is to measure zinc status and related proteins in patients with Thalassemia who have or do not have diabetes. The secondary aim will be to explore the effect of zinc supplementation on glucose metabolism in patients with thalassemia.

DETAILED DESCRIPTION:
Patients with Thalassemia major (Thal) require frequent blood transfusions and are at risk for iron overload. High tissue iron increases the risk of various endocrinopathies, including diabetes, as well as cardiovascular disease, and infections due to the formation of free radicals. This systemic condition of oxidative stress elicits an antioxidant response to reduce tissue damage. Zinc is an important component of that response because it can compete with iron for multiple cellular binding sites and, therefore, reduce the redox-cycling of iron and minimize iron-mediated oxidation of lipids, proteins, and DNA.

In Thal patients with chronic hepatic iron overload, tissue zinc redistribution is likely to be persistent. This could create an unbalanced tissue zinc distribution with excessive amounts in the liver and deficient levels in other tissues altering zinc-dependent functions, such as growth, skeletal development, immunity, and glucose regulation. There is a rich body of literature focused on the 'diabetogenic effects' of altered zinc status which will be reviewed herein. Our group has recently shown that supplementation with 25 mg/d of zinc can improve bone density in patients with Thal. This provides evidence for a functional zinc deficiency, which may also affect other whole body zinc functions, such as insulin secretion and glucose homeostasis.

Our hypothesis is that hepatic iron overload induces a sub-clinical inflammatory response that alters the expression of MT and zinc-transport proteins leading to hepatic zinc sequestration, and an associated zinc-depletion in other tissues. Marginal zinc depletion in turn leads to increased oxidative stress, cellular apoptosis and altered glucose homeostasis and insulin secretion. This proposal will focus on cross-sectional differences in markers of glucose homeostasis and zinc status in diabetic and non-diabetic Thal patients, combined with a short- term zinc supplementation to explore the effect on glucose and insulin homeostasis.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with transfusion dependent thalassemia
* > 12 years of age

Exclusion Criteria (for both cross-sectional and interventional studies)

* patients who are pregnant
* patients who are on growth hormone therapy

Exclusion criteria (for intervention study only)

* patients who currently have diabetes (therefore cannot have an oral glucose tolerance test)

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-11; Primary Completion 2015-01 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Oral glucose Tolerance Test | 3 months
  Effect of 3 months of zinc supplementation on oral glucose tolerance test results

SECONDARY OUTCOMES:
Fructosamine | 3 months
  Determine the effect of 3 months of zinc supplementation on fructosamine levels

CONTACTS AND LOCATIONS:
Overall Officials: Ellen B Fung, PhD RD, Principal Investigator — UCSF Benioff Children's Hospital Oakland
Locations (1):
- Children's Hospital & Research Center Oakland, Oakland, California, United States